CLINICAL TRIAL: NCT03292289
Title: Assessment of Symptoms and Their Consequences on Patients Quality of Life After Coloanal Continuity Reconstruction Following a Proctectomy for Rectal Cancer
Brief Title: Assessment of Symptoms and Consequences of Coloanal Continuity Reconstruction
Acronym: QUALIPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Santelys Association (Other); Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: QUALIPRO-1703; 2017-A01406-47 (Other: ANSM)
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer
Keywords: proctectomy; coloanal continuity reconstruction
MeSH Terms: conditions — Rectal Neoplasms | interventions — Lead; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study process (Experimental): Pre- and post-operative consultations. Stomatherapy consultation. Questionnaires
  Interventions: Procedure: Pre- and post-operative consultation; Procedure: Stomatherapy consultation; Procedure: Questionnaires

INTERVENTIONS:
Procedure: Pre- and post-operative consultation — Before and between the two interventions
Procedure: Stomatherapy consultation — Clinical exam. At one and six months after the 2nd intervention
Procedure: Questionnaires — * QLQ-C30 and QLQ-CR29 at each time defined by the study (one month before and after the first intervention, before the 2nd intervention and at 1, 3, 6 and 12 months after the 2nd intervention)
  * Stoma-QoL before and after the 2nd intervention
  * LARS score at 1, 3, 6 and 12 months after the 2nd intervention

SUMMARY:
This study is a prospective, monocentric study whose aim is to assess the quality of life for patients who underwent a coloanal continuity reconstruction and to understand the functional issues they encounter. This will potentially provide predictive factors identification of bad functional outcomes allowing to guide future decisions. Also, it will allow patients to have a reinforced follow-up during the year after the reconstruction.

DETAILED DESCRIPTION:
First of all, an information document will be given to the patients and their consent will be collected. Then, they will be registered through the online eCRF (or by FAX) and a study number will be given to each patient.

The study will proceed with 2 stomatherapy consultations at one and six months after coloanal continuity reconstruction. Patient care and following up will proceed as usual. The stomatherapy consultation will be done by a qualified nurse.

Before the 1st intervention (proctectomy):

* Collect of clinical data and disease history
* Quality of life questionnaires (EORTC-QLQ-C30 and CR29)
* Evaluation of LARS score

After the 1st intervention (proctectomy, at month 1):

- Quality of life : EORTC-QLC30 and CR-29 questionnaires and Stom-QoL

Before the 2nd intervention (coloanal continuity reconstruction):

- Quality of life : EORTC-QLC30 and CR-29 questionnaires and Stom-QoL

After the 2nd intervention (at month 1, month 3, month 6 and one year):

* at 1 and 6 months : clinical exam (stomatherapy consultation) for collect of postoperative complications
* Quality of life : EORTC-QLC30 and CR-29 questionnaires and LARS score

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* Patients who are going to undergo a proctectomy for a rectal cancer (situated at a distance equal or lower to 15 cm from the anoderm) following by a coloanal continuity reconstruction (using direct, latero-terminal or colonic J-pouch anastomosis)
* Already underwent or not a neoadjuvant radio-chemotherapy
* Affiliation to the National Social Security System
* With informed and signed consent

Exclusion Criteria:

* Unwilling patients
* Patient deprived of their liberty or under guardianship or tutorship.
* Abdominal perineal amputation
* No stoma placement planned
* Tumor more than 15 cm from the anal margin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Quality of life 1 year after the second intervention, using LARS score | from baseline to 1 year after the second intervention
  Obtain an objective assessment of symptoms intensity (using the LARS score)for patients who received a proctectomy for rectal cancer ("1st intervention") following by a coloanal continuity reconstruction ("2nd intervention")

SECONDARY OUTCOMES:
Quality of life before the first intervention and after the second intervention | from baseline to one year after the 2nd intervention
  Obtain an objective assessment of symptoms intensity (using the LARS score)for patients who received a proctectomy for rectal cancer ("1st intervention") following by a coloanal continuity reconstruction ("2nd intervention")
Quality of life using EORTC-QLQ-C30 | from baseline to one year after the 2nd intervention
  Assess the quality of life using EORTC-QLQ-C30 questionnaires before the first intervention, between the first and the second intervention and after the second intervention
Quality of life using EORTC-QLQ-CR29 questionnaires | from baseline to one year after the 2nd intervention
  Assess the quality of life using EORTC-QLQ- CR29 questionnaires before the first intervention, between the first and the second intervention and after the second intervention
Impact of stomy on quality of life | from the first intervention to 6 months after the first intervention
  Assess the impact of stomy on quality of life for patients who received a proctectomy for rectal cancer and using Stoma-QoL questionnaire
Rate of patients with anastomotic fistula | from the first intervention to 6 months after the first intervention
  Determinate the rate of patients with anastomotic fistula requiring the conservation of the stomy, and so they cannot undergo a coloanal continuity reconstruction
Surgical complications description | from first intervention to one year after the 2nd intervention
  Describe surgical complications linked to the coloanal continuity reconstruction
Quality of life of patients with a second stoma placement, using EORTC-QLQ-CR29 questionnaires | From the 2nd intervention to one year after the 2nd intervention
  Assess the quality of life of patients who have a new stoma for functional disorder after restoration of digestive continuity .
Quality of life of patients with a second stoma placement, using EORTC-QLQ-C30 questionnaires | From the 2nd intervention to one year after the 2nd intervention
  Assess the quality of life of patients who have a new stoma for functional disorder after restoration of digestive continuity .
Quality of life of patients with a second stoma placement, using LARS score | From the 2nd intervention to one year after the 2nd intervention
  Assess the quality of life of patients who have a new stoma for functional disorder after restoration of digestive continuity .

CONTACTS AND LOCATIONS:
Overall Officials: Pascale COULON, Study Director — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No